CLINICAL TRIAL: NCT05152667
Title: Ambispective Comparative Cohort Study to Assess the Effect of Pretreatment With a Levonorgestrel-Releasing Intrauterine System Versus Oral Progestin on ICSI and Vitrified-Warmed Embryo Transfer Outcomes in Women With Adenomyosis
Brief Title: Ambispective Study to Assess the Effect of Pretreatment With a Levonorgestrel-Releasing Intrauterine System Versus Oral Progestin
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wael Elbanna Clinic (Other)
Collaborators: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Wael Elbanna, Managing director for Wael Elbanna Clinic, Wael Elbanna Clinic
Other Study IDs: Elbanna_001
Record Dates: First submitted 2021-08-13; First posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-08

CONDITIONS: Adenomyosis; IVF
MeSH Terms: conditions — Adenomyosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm 1: Women with adenomyosis pretreated with levonorgestrel-releasing intrauterine device (LNG-IUS) and proceeding with the ICSI
  Interventions: Device: levonorgestrel-releasing intrauterine device (LNG-IUS)
- Arm 2: Women with adenomyosis pretreated with oral progestin "Dienogest" and proceeding with the ICSI

INTERVENTIONS:
Device: levonorgestrel-releasing intrauterine device (LNG-IUS) — Intervention is administered proceeding the ICSI
  Other Names: oral progestin "Dienogest"
  Groups: Arm 1

SUMMARY:
The study participants' relevant medical records will be collected and reviewed for the retrospective subjects and after obtaining informed consent for the prospective subjects. The study materials that will be used will include blood tests, transvaginal ultrasound and magnetic resonance imaging (MRI). The study will involve two study arms

DETAILED DESCRIPTION:
The study participants' relevant medical records will be collected and reviewed for the retrospective subjects and after obtaining informed consent for the prospective subjects. The study materials that will be used will include blood tests, transvaginal ultrasound and magnetic resonance imaging (MRI). The study will involve two study arms:

Arm 1: Women with adenomyosis pretreated with levonorgestrel-releasing intrauterine device (LNG-IUS) and proceeding with the ICSI Arm 2: Women with adenomyosis pretreated with oral progestin "Dienogest" and proceeding with the ICSI Primary and secondary key measurements will be used in the study.

The primary measures will include:

* Presence of intrauterine gestational sac at 12 weeks
* Presence of fetal heart pulsation at 12 weeks

The secondary key measures will include:

* Occurance of abortion in the 1st trimester
* Appearance of ectopic pregnancy diagnosis by:

Ultrasound Serum β-HCG level Symptoms of pain and bleeding

* Two serum β-HCG levels in 48hrs interval to emphasis biochemical pregnancy
* Recording the the baseline characteristics of the study participants

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed using both the transvaginal ultrasound study (TVS) and MRI criteria

   * Main criteria for sonographic and MRI diagnosis of adenomyosis are:

   The appearance of asymmetrical thickening of the myometrium Irregular cystic areas within the myometrium Linear striations radiating out from the myometrium
2. Patients ≤42 years old at the time of starting ICSI cycle
3. Cryopreserved embryo transfer cycles
4. The presence of at least one good cryopreserved day 3 embryo.

Exclusion Criteria:

1. Transfer of a poor-quality embryo (grades 3 or 4)
2. History of myomectomy
3. Pelvic ultrasound that showed the presence of uterine fibroids, a hydrosalpinx or endometrial polyps (all known causes of implantation failure).

Max Age: 42 Years | Sex: Female
Age Groups: Child, Adult
Gender Based: Yes
Study Population: The study population will include women with adenomyosis, proceeding with the ICSI and pretreated with either:
  1. levonorgestrel-releasing intrauterine device (LNG-IUS)
  2. Oral progestin "Dienogest"
Sampling Method: Non-Probability Sample
Enrollment: 354 (Estimated)
Dates: Start 2021-11-27 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
ongoing pregnancy | up to 13 weeks gestation
  - Recording the following for the two arms of the study: Presence of intrauterine gestational sac at 12 weeks Presence of fetal heart pulsation at 12 weeks

SECONDARY OUTCOMES:
Occurance of abortion or ectopic | up to 13 weeks gestation
  Recording the following for the two arms of the study:
  Occurance of abortion in the 1st trimester Appearance of ectopic pregnancy diagnosis Two serum β-HCG levels in 48hrs interval
Recording the baseline characteristics of the study participants | Before study intervention
  age
Recording the baseline characteristics of the study participants | Before study intervention
  BMI in kg/m^2

CONTACTS AND LOCATIONS:
Locations (1):
- Wael Elbanna Clinic, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided